CLINICAL TRIAL: NCT00425620
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Group Study of Intranasal Amphotericin B Suspension in Patients With Refractory, Postsurgical Chronic Sinusitis (CS)
Brief Title: Amphotericin B Suspension in Refractory Chronic Sinusitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Accentia Biopharmaceuticals (Industry)
Responsible Party: Ben McOmber, MPH, Accentia Biopharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACC-05-01
Record Dates: First submitted 2007-01-19; First posted 2007-01-23 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Chronic Sinusitis
Keywords: Chronic Sinusitis; Chronic Rhinosinusitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amphotericin B (Experimental)
  Interventions: Drug: SinuNase

INTERVENTIONS:
Drug: SinuNase — Lavage
  Other Names: Amphotericin B Suspension

SUMMARY:
The primary objective of the study is to evaluate the safety and efficacy of Amphotericin B suspension versus placebo in the complete resolution of key chronic sinusitis symptoms during 16 weeks of treatment in patients with refractory, postsurgical CS.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of refractory, postsurgical chronic sinusitis
* Has a documented history of chronic sinusitis symptoms for more than 12 weeks
* A CT scan showing a certain level of mucosal thickening in at least 1 maxillary sinus
* An endoscopy documenting the presence of inflammation and absence of stage 4 polyps
* Ability to comply with the study requirements including the ability to administer a nasal lavage twice daily for 4 months
* Females of childbearing potential must use adequate birth control methods and not plan to get pregnant during the course of the study.
* Ability to read or speak English

Exclusion Criteria:

* Has a hypersensitivity to Amphotericin B or the compounds of any study medications
* Is an immunosuppressed patient or is receiving disease modifying agents
* Has an acute upper or lower respiratory illness
* Has an acute exacerbation of chronic sinusitis within 1 month prior to randomization
* Has used systemic antibiotic therapy for reasons other than acute sinusitis within 3 weeks prior to randomization
* Has used any antibiotic therapy for acute complication of chronic sinusitis within 1 month prior to randomization
* Has orbital or central nervous system complications
* Has acute asthma at study initiation
* Began using nasal corticosteroids or had a dosage change within 3 months prior to randomization
* Has taken a dose of oral or intravenous steroids to treat any condition other than asthma within 1 month prior to randomization
* Has used any systemic antifungal therapy within 3 months prior to randomization
* Has used intranasal antifungal therapy for chronic sinusitis within 3 months prior to randomization
* Currently has a clinically significant deviated nasal septum that has not been remedied by surgery
* Has an anatomical abnormality which would significantly obstruct the nasal passages
* Has cystic fibrosis
* Is pregnant
* Has stage 4 polyposis
* Has any significant medical condition that in a doctor's opinion could affect the patient's participation in the trial
* Has used any investigational product within 1 month of study initiation
* Has a history of cancer other than treated squamous cell or basal cell carcinoma of the skin that has not been in full remission for at least 5 years prior to study initiation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-12; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the safety and efficacy of Amphotericin B suspension versus placebo in the complete resolution of key chronic sinusitis symptoms during 16 weeks of treatment in patients with refractory, postsurgical CS. | Four months

CONTACTS AND LOCATIONS:
Overall Officials: Angelos M Stergiou, MD, Study Director — Accentia Biopharmaceuticals
Locations (68):
- United States (68):
  - Parkway Medical Center, Birmingham, Alabama
  - Alabama ENT Associates, Birmingham, Alabama
  - Clinical Research Advantage, Gilbert, Arizona
  - NEA Clinic, Jonesboro, Arkansas
  - Kern Allergy Medical Clinic, Bakersfield, California
  - SARC Research Center, Fresno, California
  - California Allergy & Asthma Medical Group, Inc., Los Angeles, California
  - CHOC PSF, AMC, Division of Allergy, Asthma & Immunology, Orange, California
  - Integrated Research Group Inc., Riverside, California
  - Allergy Medical Group of the North Area, Roseville, California
  - Sacramento ENT, Sacramento, California
  - Allergy & Asthma Clinical Research, Inc., Walnut Creek, California
  - Pravin K. Muniyappa, MD, Inc., West Hills, California
  - First Allergy & Clinical Research Center, Centennial, Colorado
  - Colorado Otolaryngology Associates, PC, Colorado Springs, Colorado
  - Connecticut Sinus Center, Bridgeport, Connecticut
  - Bay Front Medical Center, St. Petersburg, Florida
  - Allergy Center at Brookstone, Columbus, Georgia
  - Allergy & Asthma Care Center, Gainesville, Georgia
  - Northeast Georgia Research Center, Gainesville, Georgia
  - Northwest ENT Associates, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Chest Medicine Consultants, Chicago, Illinois
  - Asthma And Allergy Center Of Chicago, River Forest, Illinois
  - South Bend Clinic, South Bend, Indiana
  - Kansas City Allergy & Asthma, Overland Park, Kansas
  - Commonwealth ENT, Head and Neck Center, Louisville, Kentucky
  - Paul A. Shapero, MD, Bangor, Maine
  - Institute of Allergy & Asthma, Wheaton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hurley Medical Center, Flint, Michigan
  - Grand Traverse Allergy, Traverse City, Michigan
  - Clinical Research Institute, Plymouth, Minnesota
  - Jefferson City Medical Group, Jefferson City, Missouri
  - St. Louis University, St Louis, Missouri
  - Midwest Clinical Research, LLC, St Louis, Missouri
  - Allergy & Asthma Consultants of Montana, Bozeman, Montana
  - Central Jersey Health Care, Elizabeth, New Jersey
  - David Sherris, M.D., Buffalo, New York
  - Health Sciences Research Center, Ithaca, New York
  - Wellington Tichenor, MD, New York, New York
  - DiGiovanna Family Care Center, North Massapequa, New York
  - AAIR Research Center, Rochester, New York
  - Center for Allergy & Asthma of Bronx & Westchester, The Bronx, New York
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - Charlotte Eye, Ear, Nose & Throat Associates, P.A., Charlotte, North Carolina
  - Dr. Ann Bogard Private Practice, Winston-Salem, North Carolina
  - Odyssey Research, Bismarck, North Dakota
  - Center for Specialty Care, Fargo, North Dakota
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Optimed Research, Columbus, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - COR Clinical Research, Oklahoma City, Oklahoma
  - Allergy and Asthma Research of NJ, Inc., Philadelphia, Pennsylvania
  - ADAC Research, Greenville, South Carolina
  - Sterling ENT / Carolina Research, Orangeburg, South Carolina
  - The Asthma Institute, PLLC, Chattanooga, Tennessee
  - Jackson Clinic, Jackson, Tennessee
  - Vanderbilt University ASAP Research, Nashville, Tennessee
  - Texas Medical and Surgical Associates, Dallas, Texas
  - University Of North Texas Health Science Center, Fort Worth, Texas
  - Allergy & Asthma Associates, Houston, Texas
  - San Antonio Ear, Nose & Throat Research, San Antonio, Texas
  - Live Oak Allergy & Asthma Clinic, San Antonio, Texas
  - King's Daughters Clinic, Temple, Texas
  - Virginia Adult & Pediatric Allergy & Asthma, P.C., Richmond, Virginia
  - Liberty Research Center, Tacoma, Washington
  - Monroe Medical Foundation, Monroe, Wisconsin